CLINICAL TRIAL: NCT03475433
Title: An Observational Prospective Cohort Study About Quality of Life in Relation to the Physical Activity of Taiwanese Breast and Prostate Cancer Patients.
Brief Title: An Observational Prospective Cohort Study Using an Actigraphy Device.
Status: Completed | Type: Observational
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); University of Seville (Other); Taipei Medical University WanFang Hospital (Other); Taipei Medical University Hospital (Other); Adhera Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: None yet
Record Dates: First submitted 2018-03-05; First posted 2018-03-23 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2018-03

CONDITIONS: Neoplasm of Breast (Disorder); Carcinoma of Prostate (Disorder)
Keywords: Cancer; Questionnaire; Survey; Sleep Disturbance; Sleep Quality; E-health; M-health; Actigraphy; Physical activity; Dyssomnias Medical Subject Headings [MeSH]; Sleep Wake Disorders [MeSH]; Parasomnias [MeSH]; Nervous System Diseases [MeSH]; Mental Disorders [MeSH]; Neurologic Manifestations [MeSH]; Signs and Symptoms [MeSH]; Telemedicine [MeSH]; Actigraphy [MeSH]; Quality of Life [MeSH]; Motor Activity [MeSH]; Breast Neoplasms [MeSH]; Prostatic Neoplasms [MeSH]; Sleep Hygiene [MeSH]; Neoplasms [MeSH]
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplasms; Parasomnias; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Beast cancer patients: All participants that suffer from breast cancer.
  Interventions: Device: Actigraphy device
- Prostate cancer patients: All participants that suffer from prostate cancer.
  Interventions: Device: Actigraphy device

INTERVENTIONS:
Device: Actigraphy device — Both groups will receive an actigraphy device that will passively measure their movement data.

SUMMARY:
This study focuses on whether or not physical activity and sleep quality correlate with the health of prostate and breast cancer patients. The activity data will be acquired using wearable actigraphy devices, which the subjects will wear for the duration of seven days. The sleep quality will be measured using a combination of actigraphy and the mandarin version of the Pittsburgh Sleep Quality Index (PSQI) and the Quality of Life Questionnaire (QLQ). By using this combination, the investigators will not only measure the objective physical activity while the patient is asleep, but also the subjective sleep quality. The questionnaire will also function as control data for the accuracy of the actigraphy device.

This study will recruit approximately 30 breast or prostate cancer patients. The participants will wear a wearable actigraphy device for 7 consecutive days, which will provide accurate and objective movement and sleep data. This data is linked to a unique Identification number (ID), which will be noted in the participant's case report. This case report also contains the participant's information and answers to the questionnaires.

DETAILED DESCRIPTION:
Physical inactivity is a common issue amongst breast cancer patients. Previous studies have shown that physical activity can be beneficiary to both the cancer outcomes and the quality of life.

However, most comparable studies had western populations or included some participants of Asian descent at best. Given the growing importance of effective and efficient follow-up care [1] and the lack of research on physical activity and sleep quality in relation to the Quality of Life (QoL) of cancer patients in Asian countries, the investigators aim to monitor the physical activity, sleep quality and subjective QoL of Taiwanese breast- and prostate cancer patients. Hence the investigators' main research question is: "Does physical and/or sleep activity affect the quality of life of (Taiwanese) breast and prostate cancer patients?". If this would be the case, the results might cover the bases for an intervention study aimed at improving physical and/or sleep quality in these cancer patients.

This study focuses on whether or not physical activity and sleep quality correlate with the health of prostate and breast cancer patients. The activity data will be acquired using wearable actigraphy devices, which the subjects will wear for the duration of seven days. The sleep quality will be measured using a combination of actigraphy and the mandarin version of the Pittsburgh Sleep Quality Index (PSQI). By using this combination, the investigators will not only measure the objective physical activity while the patient is asleep, but also the subjective sleep quality. The questionnaire will also function as control data for the accuracy of the actigraphy device.

Lastly, the quality of life will be measured using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire 30 (EORTC QLQ-C30). This will provide an insight in the quality of life of the subjects, which will enable the investigators to draw a conclusion whether or not physical activity and sleep quality are related to the quality of life.

This study will recruit approximately 30 breast or prostate cancer patients. The participants will wear a wearable actigraphy device for 7 consecutive days, which will provide accurate and objective movement and sleep data. This data is linked to a unique ID, which will be noted in the participant's case report. This case report also contains the participant's information and answers to the questionnaires.

To retrieve results from the dataset, the data analysis will be divided in two parts: correlation between sleep quality and the Quality of Life, and between physical activity and the Quality of Life. Before commencing with the analysis itself, the data will be checked for outliers and missing data.

ELIGIBILITY:
Inclusion Criteria:

The patient:

* Is an outpatient receiving evaluation, treatment, or follow-up care at either one of the desired hospital locations in Taipei.
* Has been diagnosed with prostate or breast cancer within the past year.
* Is currently receiving treatment for the cancer.
* Is at least 20 years old.
* Is able to understand Mandarin Chinese.
* Gives informed consent to participate.
* scores at least 26 on the Mini-Mental State Examination (MMSE).
* Has a score 45 or higher on the Berg Balance Scale test.

Exclusion Criteria:

The patient:

* Cannot understand the intent of the study.
* scores lower than 26 on the Mini-Mental State Examination (MMSE).
* Is not fit to participate, as believed by their current treating physician.
* Is physical unable to walk.
* Has a score of <45 on the Berg Balance Scale test.
* Refuses to participate.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be selected with the help of oncologists in Taiwanese hospitals, therefore all participants will be Taiwanese residents and patients of either one of the desired hospital locations in Taipei. All participants are also either breast cancer or prostate cancer patients, with a minimum age of 20 years.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change will be assessed on the quality of life of breast and prostate cancer patients. | The time frame will be 8th day after enrolment of each respondent
  It will be measured using the scores of the Quality of Life questionnaire.
Change will be assessed for the influence of physical activity on the Quality of Life of breast and prostate cancer patients. | The time frame will be daily for 8 days after enrolment of each respondent
  It will be measured using the physical activity data from the actigraphy device.

SECONDARY OUTCOMES:
Study whether sleep quality and the quality of life scores of breast and prostate cancer patients are correlated | The time frame will be 8th day after enrollment of each respondent
  This will be measured using a combination of the PSQI questionnaire and movement data during nighttime for the sleep quality, and the quality of life questionnaire scores.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Abdul Shabbir, Dr. MD, Principal Investigator — Associate Professor & Health IT Consultant
Locations (2):
- Taiwan (2):
  - Taipei Medical University Hospital, Taipei, Taipei City
  - Taipei Municipal Wanfang Hospital, Taipei, Taipei City

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data (IPD) will be shared as open research data after the results have been published. All data that might identify individuals will be stripped to make sure the data is completely anonymous.
Supporting Information: Study Protocol
Time Frame: The anonymous (raw) data might be shared after the study itself has been finished.
Access Criteria: The applications for IPD sharing will be reviewed on an individual basis by the Principal Investigator.

REFERENCES:
- [Background] Robison LL, Demark-Wahnefried W. Cancer survivorship: focusing on future research opportunities. Cancer Epidemiol Biomarkers Prev. 2011 Oct;20(10):1994-5. doi: 10.1158/1055-9965.EPI-11-0837. No abstract available. PMID 21980006
- [Background] Monga U, Kerrigan AJ, Thornby J, Monga TN. Prospective study of fatigue in localized prostate cancer patients undergoing radiotherapy. Radiat Oncol Investig. 1999;7(3):178-85. doi: 10.1002/(SICI)1520-6823(1999)7:33.0.CO;2-0. PMID 10406060
- [Background] Shin WK, Song S, Jung SY, Lee E, Kim Z, Moon HG, Noh DY, Lee JE. The association between physical activity and health-related quality of life among breast cancer survivors. Health Qual Life Outcomes. 2017 Jun 30;15(1):132. doi: 10.1186/s12955-017-0706-9. PMID 28666465
- [Background] Inbar C, Ety B, Ayala H, Tamer P. The mental health of breast cancer survivors and their adolescent daughters. Psychooncology. 2013 Jun;22(6):1236-41. doi: 10.1002/pon.3127. Epub 2012 Jul 4. PMID 22764063
- [Background] Toivonen KI, Tamagawa R, Speca M, Stephen J, Carlson LE. Open to Exploration? Association of Personality Factors With Complementary Therapy Use After Breast Cancer Treatment. Integr Cancer Ther. 2018 Sep;17(3):785-792. doi: 10.1177/1534735417753539. Epub 2018 Jan 24. PMID 29361852
- [Background] Szymlek-Gay EA, Richards R, Egan R. Physical activity among cancer survivors: a literature review. N Z Med J. 2011 Jun 24;124(1337):77-89. PMID 21946880
- [Background] Speck RM, Courneya KS, Masse LC, Duval S, Schmitz KH. An update of controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. J Cancer Surviv. 2010 Jun;4(2):87-100. doi: 10.1007/s11764-009-0110-5. Epub 2010 Jan 6. PMID 20052559
- [Background] Meneses-Echavez JF, Gonzalez-Jimenez E, Ramirez-Velez R. Supervised exercise reduces cancer-related fatigue: a systematic review. J Physiother. 2015 Jan;61(1):3-9. doi: 10.1016/j.jphys.2014.08.019. Epub 2014 Dec 13. PMID 25511250
- [Background] Fortner BV, Stepanski EJ, Wang SC, Kasprowicz S, Durrence HH. Sleep and quality of life in breast cancer patients. J Pain Symptom Manage. 2002 Nov;24(5):471-80. doi: 10.1016/s0885-3924(02)00500-6. PMID 12547047
- [Background] Costa AR, Fontes F, Pereira S, Goncalves M, Azevedo A, Lunet N. Impact of breast cancer treatments on sleep disturbances - A systematic review. Breast. 2014 Dec;23(6):697-709. doi: 10.1016/j.breast.2014.09.003. Epub 2014 Oct 11. PMID 25307946
- [Background] Tsai PS, Wang SY, Wang MY, Su CT, Yang TT, Huang CJ, Fang SC. Psychometric evaluation of the Chinese version of the Pittsburgh Sleep Quality Index (CPSQI) in primary insomnia and control subjects. Qual Life Res. 2005 Oct;14(8):1943-52. doi: 10.1007/s11136-005-4346-x. PMID 16155782
- [Background] Wan C, Meng Q, Yang Z, Tu X, Feng C, Tang X, Zhang C. Validation of the simplified Chinese version of EORTC QLQ-C30 from the measurements of five types of inpatients with cancer. Ann Oncol. 2008 Dec;19(12):2053-60. doi: 10.1093/annonc/mdn417. Epub 2008 Jul 24. PMID 18653703
- See also: The website of the CATCH project — http://www.catchitn.eu
- See also: Information about our research facility — http://ichit.tmu.edu.tw